CLINICAL TRIAL: NCT05490784
Title: Effects of Lee Silverman Voice Treatment BIG on Dynamic Balance in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0253
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease; Motor Disorders; Balance; Distorted
Keywords: Parkinson Disease; Balance; Distorted; Motor Disorders
MeSH Terms: conditions — Parkinson Disease; Motor Disorders

STUDY DESIGN:
Intervention Model Description: total 26 participants will be randomly assigned to experimental group (Lee Silverman Voice Treatment BIG along with conventional therapy) and control group( conventional treatment)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lee Silverman Voice Treatment big with conventional treatment (Experimental): Lee Silverman Voice Treatment big with conventional treatment
  Interventions: Other: Lee Silverman Voice Treatment BIG
- control group (Active Comparator): Patients assigned to control group received conventional treatment program encompassing set of exercises such as complex motor sequences, stretching, dual tasking, mental imagery and core stability.
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Lee Silverman Voice Treatment BIG — Patients assigned to experimental group will get Lee Silverman Voice Treatment BIG along with conventional treatment.
  Arms: Lee Silverman Voice Treatment big with conventional treatment
Other: conventional treatment — patients in this group will get conventional treatment program encompassing set of exercises such as complex motor sequences, stretching, dual tasking, mental imagery and core stability.
  Arms: control group

SUMMARY:
To determine the effects of Lee Silverman Voice Treatment BIG on dynamic balance in Parkinson's patients

DETAILED DESCRIPTION:
This study will be conducted to compare the effects of Lee Silverman Voice Treatment BIG and conventional physiotherapy on dynamic balance in patients of PD. Patients will be recruited according to inclusion criteria and data will be collected from Riphah rehabilitation center, National Hospital Lahore. Dynamic gait index will be used as data collection tool to test dynamic balance of patients. Patients will be allocated to intervention groups by randomization. After approval from ethical committee, data collection will be started and informed consent will be taken from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage I, II, III Parkinson's patients on Hoehn &;Yahr classification
* Able to walk without assistive devices
* Stable medication 4 weeks prior to and during study

Exclusion Criteria:

* Patients with depression or dementia
* Disabling bradykinesia to make sure patients are efficient to engage and cooperate in conventional physical therapy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | 9 months
  Dynamic gait index assesses postural stability, gait, and balance. It evaluates various gait- related tasks with challenging situations such as head turn, speed change, obstacles and stairs climbing.

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oguz S, Erturk G, Polat MG, Apaydin H. The effect of kinesiophobia on physical activity, balance, and fear of falling in patients with Parkinson's disease. Physiother Theory Pract. 2023 Apr;39(4):865-872. doi: 10.1080/09593985.2022.2028325. Epub 2022 Jan 18. PMID 35042438
- [Background] Fleming Walsh S, Balster C, Chandler A, Brown J, Boehler M, O'Rear S. LSVT BIG(R) and long-term retention of functional gains in individuals with Parkinson's disease. Physiother Theory Pract. 2022 May;38(5):629-636. doi: 10.1080/09593985.2020.1780655. Epub 2020 Jun 17. PMID 33969801
- [Background] Schaible F, Maier F, Buchwitz TM, Schwartz F, Hoock M, Schonau E, Libuda M, Hordt A, van Eimeren T, Timmermann L, Eggers C. Effects of Lee Silverman Voice Treatment BIG and conventional physiotherapy on non-motor and motor symptoms in Parkinson's disease: a randomized controlled study comparing three exercise models. Ther Adv Neurol Disord. 2021 Feb 18;14:1756286420986744. doi: 10.1177/1756286420986744. eCollection 2021. PMID 33680093
- [Background] Tremblay C, Abbasi N, Zeighami Y, Yau Y, Dadar M, Rahayel S, Dagher A. Sex effects on brain structure in de novo Parkinson's disease: a multimodal neuroimaging study. Brain. 2020 Oct 1;143(10):3052-3066. doi: 10.1093/brain/awaa234. PMID 32980872